CLINICAL TRIAL: NCT02109939
Title: 12 Week, Randomized, Double-Blind, Controlled Evaluation Followed by an Open Label 12-Week Follow-up Period of the Impact of GeneSight Psychotropic on Response to Psychotropic Treatment in Outpatients Suffering From A Major Depressive Disorder (MDD) Having Had- Within the Current Episode- An Inadequate Response to at Least One Medication Included in GeneSight Psychotropic
Brief Title: Genomics Used to Improve DEpression Decisions
Acronym: GUIDED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assurex Health Inc. (Industry)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARX1006
Record Dates: First submitted 2014-04-04; First posted 2014-04-10 (Estimated); Results first posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: MDD; Pharmacogenomic; Pharmacogenomic Testing; Pharmacogenomics; Genetic Testing; Genetics; Major Depressive Disorder; GeneSight; Assurex; AssureRx; Psychotropic; Randomized; Double Blind; Placebo Controlled
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GeneSight Psychotropic Tested (Active Comparator): Subjects being tested with GeneSight Psychotropic
  Interventions: Genetic: GeneSight Psychotropic
- Treatment As Usual (Placebo Comparator): This group of subjects will not see their GeneSIght results or know whether or not they are in either arm until after week 12.
  Interventions: Genetic: GeneSight Psychotropic

INTERVENTIONS:
Genetic: GeneSight Psychotropic — The GeneSight Psychotropic product is a pharmacogenomic decision support tool that helps clinicians to make informed, evidence-based decisions about proper drug selection, based on the testing for clinically important genetic variants in multiple pharmacokinetic and pharmacodynamic genes that affect a patient's ability to tolerate or respond to medications.
  The GeneSight Psychotropic product contains the most commonly prescribed antidepressant and antipsychotic medications, including a full representation of the SSRI and SNRI drug classes.
  tricyclic antidepressants, an MAOI, and typical and atypical antipsychotics are also represented.
  Other Names: Assurex Health; GeneSight

SUMMARY:
Evaluate the impact of GeneSight Psychotropic on response to psychotropic treatment as judged by the mean change in the 17-item Hamilton Depression (HAM-D17) score from baseline to end of Week 8 of the study.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a highly prevalent (Hasin et al., 2005) mental disorder and a leading source of disease burden worldwide (Lopez et al., 2006). Epidemiological studies estimate 12-month and lifetime prevalence for MDD in the United States to be 5.3% and 13.2%, respectively (reviewed in Blanco et al., 2010). MDD is expected to be the second greatest cause of disability by 2020 and has been shown to cause significant morbidity, affecting people's ability to work, function in relationships, and engage in social activities. Moreover, MDD increases the risk of suicidal ideation, attempted suicide, and death by completed suicide.

Prospective longitudinal studies of patient samples show that MDD is a chronic illness, characterized by remitting and recurrent depressive episodes (Solomon et al., 1997; Mueller et al., 1999). A major depressive episode is characterized by a low mood or an inability to experience pleasure (anhedonia), or both, for more than 2 weeks, combined with several cognitive and vegetative symptoms and the occurrence of distress or impairment (reviewed in Rot et al., 2009). In the US, nearly 1 in 5 people will experience a major depressive episode at some point in their lives (reviewed in Rot et al., 2009). Drugs currently available to treat depression fall into the categories of those that have their main effect by increasing norepinephrine (NE) (the tricyclic or tetracyclic antidepressants [TCAs]), those that increase serotonin (5-HT) (the selective serotonin reuptake inhibitors [SSRIs]), and those that increase both NE and 5-HT (the monoamine oxidase inhibitors [MAOIs] and the serotonin and norepinephrine reuptake inhibitors [SNRIs]). While all antidepressants achieve similar levels of efficacy, treatment failures are relatively high ranging from 30 to 60% (Simpson and DePaulo). Additionally, many of these compounds are associated with significant adverse events (AEs).

The GeneSight Psychotropic product is a pharmacogenomic decision support tool that helps clinicians to make informed, evidence-based decisions about proper drug selection, based on the testing for clinically important genetic variants in multiple pharmacokinetic and pharmacodynamic genes that affect a patient's ability to tolerate or respond to medications.

The GeneSight Psychotropic product contains the most commonly prescribed antidepressant and antipsychotic medications, including a full representation of the SSRI and SNRI drug classes.

Tricyclic antidepressants, an MAOI, and typical and atypical antipsychotics are also represented.

The clinical utility of GeneSight Psychotropic has been evaluated in three previous prospective trials. Hall-Flavin et al reported the results of an open-label pilot study (n = 44) comparing GeneSight guided treatment to treatment as usual (TAU) without the benefit of pharmacogenomic testing (2012). The GeneSight guided arm demonstrated a 30.8% improvement in HAM-D17 score by the end of the 8 week treatment period, compared to an 18.2% improvement in the TAU arm (p = 0.04). Results of the larger (n = 165) open-label trial (Hall-Flavin, et al 2013) mirrored these findings, demonstrating a 46.9% improvement in HAMD17 score in the GeneSight arm, compared to a 29.9% improvement in the TAU arm (p < 0.0001). The third trial used a randomized, double-blind trial design (n = 51). Due to the small sample size, the trial was underpowered to detect a significant difference in improvement between the two arms (TAU and GeneSight). However, effect sizes of improvement reflected those seen in previous trials. The GeneSight group experienced a 30.8% improvement in HAMD17, compared to 20.7% in TAU. Odds ratios for response were calculated, showing that GeneSight-guided subjects had a 2.14 times greater likelihood of response compared to TAU subjects, which was similar to the 4.67 (smaller trial) and 2.06 (larger trial) odds ratios calculated for the other two studies.

Previous studies utilizing an open-label design have shown significant improvement in patient outcomes following use of the GeneSight test. However, although effect sizes were similar to those seen in the open-label studies, a small (n = 51) blinded, randomized controlled trial did not detect a statistically significant outcome. Therefore, the primary rationale for this trial is to replicate previous findings of improvement in clinical outcomes in subjects treated with the benefit of GeneSight testing utilizing a double-blind, randomized control trial (RCT) design.

It is expected that results from this trial will be used to inform guidelines for the use of pharmacogenomic testing for the treatment of major depressive disorder. Results may also be shared with regulatory bodies in the United States and abroad.

ELIGIBILITY:
Inclusion Criteria:

* Be able to understand the requirements of the study and provide written informed consent to participate in this study; a signed and dated ICF will be obtained from each patient before participation in the study;
* Have provided written authorization for the use and disclosure of their protected health information;
* Be ≥18 years of age;
* Suffer from a Major Depressive Episode meeting DSM-IV-TR criteria;
* Have had an inadequate response within the current episode to at least 1 psychotropic treatment. Inadequate response is defined as inadequate efficacy after 6 weeks of a psychotropic treatment or discontinuation of a psychotropic treatment due to AEs or intolerability;
* Have a total baseline score on the QIDS-C16 and QIDS-SR16 rating scale ≥11;
* Agree to abide by the study protocol and its restrictions and be able to complete all aspects of the study, including all visits and tests.

Exclusion Criteria:

* Patients posing a serious suicidal risk and/or in need of immediate hospitalization as judged by the investigator;
* Patients with a diagnosis of Bipolar I or II disorder;
* Patients with a current Axis I diagnosis of:

  1. Delirium
  2. Dementia
  3. Amnestic and other cognitive disorder
  4. Schizophrenia or other psychotic disorder;
* Patients having experienced hallucinations, delusions, or any psychotic symptomatology within the current depressive episode or during prior depressive episodes;
* Patient is currently in an inpatient facility;
* Patients with a history of hypothyroidism unless taking a stable dose of thyroid medication and asymptomatic or euthyroid for 6 months;
* Patients who meet DSM-IV-TR criteria for any significant current substance use disorder;
* Patients with significant unstable medical condition; life threatening disease; hepatic insufficiency (3X ULN for AST and/or ALT); liver transplant recipient; cirrhosis of the liver; need for therapies that may obscure the results of treatment and/or of the study; malignancy (except basal cell carcinoma) and/or chemotherapy within 1 year prior to screening; malignancy more than 1 year prior to screening must have been local and without metastasis and/or recurrence, and if treated with chemotherapy, without nervous system complications;
* Participation in another clinical trial within 30 days of the screening visit;
* Anticipated inability to attend scheduled study visits;
* Patients who in the judgment of the Investigator may be unreliable or uncooperative with the evaluation procedure outlined in this protocol;
* Patients with a history of prior pharmacogenomic testing;
* Any change in psychotropic medication (including change in dosage) between screening and randomization;
* Patients receiving ECT, DBS or TMS treatment (should a Subject receive any of these treatments they must be discontinued from the study);
* Patients who are known to be pregnant or lactating;
* Patients with a history of gastric bypass surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1398 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Greden, Ph.D, Principal Investigator — University of Michigan
Locations (61):
- United States (61):
  - Birmingham Psychiatry Pharmaceutical Studies, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - CiTrials, Bellflower, California
  - Catalina Research Institute, Chino, California
  - CiTrials, Costa Mesa, California
  - Synergy Research Center, Escondido, California
  - Pharmacology Research Institute, Los Alamitos, California
  - North County Research, Oceanside, California
  - CiTrials, Riverside, California
  - Stanford School of Medicine, Stanford, California
  - Viking Clinical Research, Temecula, California
  - Elite Clinical Trials, Inc, Wildomar, California
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - Howard University Hospital Mental Health Clinic, Washington D.C., District of Columbia
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions Healthcare, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Clinical Research Trials of Florida, Inc, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Janus Center For Psychiatric Research, West Palm Beach, Florida
  - Atlanta Institute of Medicine and Research, Atlanta, Georgia
  - Mood and Anxiety Program at Emory University, Atlanta, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - Carman Research, Smyrna, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Behavioral Healthcare Associates, Schaumburg, Illinois
  - The Institute of Psychiatric Research, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Kansas University Medical Center- Clinical Trials Unit, Wichita, Kansas
  - Pharmasite Research, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Geriatric Outpatient Unit- McLean Hospital, Belmont, Massachusetts
  - Boston Clinical Trials, Boston, Massachusetts
  - UMASS Center for Psychopharmacologic Research and Treatment, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - PsychCare Consultants Research, St Louis, Missouri
  - Meridian Clinical Research, Bellevue, Nebraska
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - United Medical Research Associates, Binghamton, New York
  - Integrative Clinical Trials, LLC, Brooklyn, New York
  - SPRI Clinical Trials, Brooklyn, New York
  - Eastside Comprehensive Medical Center, LLC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - University of Cincinnati Health, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Department of Psychiatry, Columbus, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Suburban Research Associates, Media, Pennsylvania
  - Mood and Anxiety Disorders Treatment and Research, Philadelphia, Pennsylvania
  - Lincoln Research, Lincoln, Rhode Island
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Alliance Research Group, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network, Seattle, Washington
  - Frontier Institute, Spokane, Washington

REFERENCES:
- [Derived] Dunlop BW, Parikh SV, Rothschild AJ, Thase ME, DeBattista C, Conway CR, Forester BP, Mondimore FM, Shelton RC, Macaluso M, Logan J, Traxler P, Li J, Johnson H, Greden JF. Comparing sensitivity to change using the 6-item versus the 17-item Hamilton depression rating scale in the GUIDED randomized controlled trial. BMC Psychiatry. 2019 Dec 27;19(1):420. doi: 10.1186/s12888-019-2410-2. PMID 31881956
- [Derived] Thase ME, Parikh SV, Rothschild AJ, Dunlop BW, DeBattista C, Conway CR, Forester BP, Mondimore FM, Shelton RC, Macaluso M, Li J, Brown K, Jablonski MR, Greden JF. Impact of Pharmacogenomics on Clinical Outcomes for Patients Taking Medications With Gene-Drug Interactions in a Randomized Controlled Trial. J Clin Psychiatry. 2019 Oct 31;80(6):19m12910. doi: 10.4088/JCP.19m12910. PMID 31721487
- [Derived] Greden JF, Parikh SV, Rothschild AJ, Thase ME, Dunlop BW, DeBattista C, Conway CR, Forester BP, Mondimore FM, Shelton RC, Macaluso M, Li J, Brown K, Gilbert A, Burns L, Jablonski MR, Dechairo B. Impact of pharmacogenomics on clinical outcomes in major depressive disorder in the GUIDED trial: A large, patient- and rater-blinded, randomized, controlled study. J Psychiatr Res. 2019 Apr;111:59-67. doi: 10.1016/j.jpsychires.2019.01.003. Epub 2019 Jan 4. PMID 30677646

RESULTS

PARTICIPANT FLOW:
Groups:
- GeneSight Psychotropic Tested: Subjects being tested with GeneSight Psychotropic
  GeneSight Psychotropic: The GeneSight Psychotropic product is a pharmacogenomic decision support tool that helps clinicians to make informed, evidence-based decisions about proper drug selection, based on the testing for clinically important genetic variants in multiple pharmacokinetic and pharmacodynamic genes that affect a patient's ability to tolerate or respond to medications.
  The GeneSight Psychotropic product contains the most commonly prescribed antidepressant and antipsychotic medications, including a full representation of the SSRI and SNRI drug classes.
  tricyclic antidepressants, an MAOI, and typical and atypical antipsychotics are also represented.
- Treatment As Usual: This group of subjects will not see their GeneSIght results or know whether or not they are in either arm.
  GeneSight Psychotropic: The GeneSight Psychotropic product is a pharmacogenomic decision support tool that helps clinicians to make informed, evidence-based decisions about proper drug selection, based on the testing for clinically important genetic variants in multiple pharmacokinetic and pharmacodynamic genes that affect a patient's ability to tolerate or respond to medications.
  The GeneSight Psychotropic product contains the most commonly prescribed antidepressant and antipsychotic medications, including a full representation of the SSRI and SNRI drug classes.
  tricyclic antidepressants, an MAOI, and typical and atypical antipsychotics are also represented.
Period: Overall Study
Arm/Group | GeneSight Psychotropic Tested | Treatment As Usual
Started | 681 | 717
Completed | 560 | 607
Not Completed | 121 | 110

BASELINE CHARACTERISTICS:
Population: Per Protocol Population at Baseline
Groups:
- Total: Total of all reporting groups
Arm/Group | GeneSight Psychotropic Tested | Treatment As Usual | Total
Number analyzed (Participants) | 681 | 717 | 1398
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 597 | 616 | 1213
  >=65 years | 84 | 101 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (14.5) | 48.0 (50.0) | 47.5 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 489 | 498 | 987
  Male | 192 | 219 | 411
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 3 | 8
  Asian | 12 | 17 | 29
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 114 | 94 | 208
  White | 538 | 589 | 1127
  More than one race | 11 | 14 | 25
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 681 | 717 | 1398
Baseline HAM-D17 [Mean (Standard Deviation); unit: units on a scale] — HAM-D17 score at baseline
  units on a scale | 21.1 (4.20) | 21.4 (4.22) | 21.3 (4.21)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the 17-item Hamilton Depression (HAM-D17) Score From Baseline to 8 Weeks
Description: Evaluate the impact of GeneSight Psychotropic on response to psychotropic treatment as judged by the mean percent change in the 17-item Hamilton Depression (HAM-D17) score from baseline to end of Week 8 of the study. Scores range from 0 to 50, and lower scores are better outcomes. Percent change is defined as (week 8 score -baseline score) / (baseline score) x 100.
Time Frame: from baseline to end of Week 8
Population: Per-Protocol
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Groups:
- Treatment As Usual: This group of subjects will not have treatment guided by their GeneSight results or know whether they are in a particular arm.
  GeneSight Psychotropic: The GeneSight Psychotropic product is a pharmacogenomic decision support tool that helps clinicians make informed, evidence-based decisions about proper drug selection, based on the testing for clinically important genetic variants in multiple pharmacokinetic and pharmacodynamic genes that affect a patient's ability to tolerate or respond to medications.
  The GeneSight Psychotropic product contains the most commonly prescribed antidepressant and antipsychotic medications, including a full representation of the SSRI and SNRI drug classes. Tricyclic antidepressants, one MAOI, and typical and atypical antipsychotics are also represented.
- GeneSight Psychotropic Tested: Subjects being tested with GeneSight Psychotropic. This group of subjects will not know whether they are in a particular arm.
  GeneSight Psychotropic: The GeneSight Psychotropic product is a pharmacogenomic decision support tool that helps clinicians make informed, evidence-based decisions about proper drug selection, based on the testing for clinically important genetic variants in multiple pharmacokinetic and pharmacodynamic genes that affect a patient's ability to tolerate or respond to medications.
  The GeneSight Psychotropic product contains the most commonly prescribed antidepressant and antipsychotic medications, including a full representation of the SSRI and SNRI drug classes. Tricyclic antidepressants, one MAOI, and typical and atypical antipsychotics are also represented.
Arm/Group | Treatment As Usual | GeneSight Psychotropic Tested
Number analyzed (Participants) | 607 | 560
percentage of change | -24.39 (1.22) | -27.23 (1.27)
Statistical Analysis 1: Comparison: Treatment As Usual vs GeneSight Psychotropic Tested; Test type: Superiority; p = 0.1070, Mixed Models Analysis; Repeated Measures including week 4; Mean Difference (Net) = -2.836, 95% CI 2-sided [-6.285 to 0.613], Standard Error of Mean 1.758

2. Secondary Outcome: Percent Change in the 16-item Quick Inventory of Depression Symptomology (QIDS-C16) Score From Baseline to 8 Weeks
Description: Mean percent change in the 16-item Quick Inventory of Depression Symptomology (QIDS-C16) score from baseline to end of Week 8 of the study. Scores range from 0 to 27 with lower scores being better outcomes. Percent change is defined as (week 8 score - baseline score) / (baseline score) x 100.
Time Frame: from baseline to end of Week 8
Population: Intent-to-Treat
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Arm/Group | GeneSight Psychotropic Tested | Treatment As Usual
Number analyzed (Participants) | 621 | 677
percentage of change | -35.107 (1.189) | -32.900 (1.147)
Statistical Analysis 1: Comparison: GeneSight Psychotropic Tested vs Treatment As Usual; Test type: Superiority; p = 0.1822, Mixed Models Analysis; MMRM with week 4 data; Mean Difference (Net) = -2.207, 95% CI 2-sided [-5.450 to 1.036], Standard Error of Mean 1.653

3. Secondary Outcome: Percentage of Responders at Week 8 for HAM-D17
Description: Adjusted percentage of responders at Week 8 in each treatment group on the 17-item Hamilton Depression Rating Scale (HAM-D17). A responder is defined as a participant with at least a 50% decrease from baseline in total scale score. Scores range from 0 to 50, and lower scores are better outcomes.
Time Frame: Week 8 visit info
Population: Per Protocol
Measure: Number; unit: percentage of subjects
Arm/Group | GeneSight Psychotropic Tested | Treatment As Usual
Number analyzed (Participants) | 560 | 607
percentage of subjects | 26.00 | 19.92
Statistical Analysis 1: Comparison: GeneSight Psychotropic Tested vs Treatment As Usual; Test type: Superiority; p = 0.0134, Generalized linear mixed model; The reported outcome measure is the estimated percentage from a generalized linear mixed model, not a simple count of subjects; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.07 to 1.86]

4. Secondary Outcome: Percentage of Responders at Week 12 for HAM-D17
Description: *Comment*: For patients in TAU, clinicians were blinded to the pharmacogenomic test result until after completion of the week 8 visit. Because unblinding might have occurred for some patients prior to week 12 assessments, data collected at week 12 were no longer considered blinded and are not analyzed or reported.
Time Frame: Week 12 visit info
Reporting Status: Not Posted

5. Secondary Outcome: Percentage of Remitters at Week 12 Defined as HAM-D17 ≤7
Description: as for outcome 4
Time Frame: week 12 visit info
Reporting Status: Not Posted

6. Secondary Outcome: Percentage of Remitters at Week 8 Defined as HAM-D17 ≤7 Each Treatment Group;
Description: Adjusted percentage of remitters at Week 8 defined as a score ≤7 in the 17-item Hamilton Depression Rating Scale (HAM-D17) in each treatment group. Scores range from 0 to 50, and lower scores are better outcomes.
Time Frame: week 8 visit info
Population: Per Protocol
Measure: Number; unit: percentage of subjects
Arm/Group | GeneSight Psychotropic Tested | Treatment As Usual
Number analyzed (Participants) | 560 | 607
percentage of subjects | 15.30 | 10.08
Statistical Analysis 1: Comparison: GeneSight Psychotropic Tested vs Treatment As Usual; Test type: Superiority; p = 0.0066, Generalized linear mixed model; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.14 to 2.27]

7. Secondary Outcome: Time to Response/Remission of Depressive Symptoms Over 8 Weeks;
Description: *Comment*: Time to response/remission is not an outcome measure that can accurately be reported from the way the data was collected. As specified in the updated SAP before the blind was broken, this was not analyzed or reported.
Time Frame: week 4 and 8 visit info
Reporting Status: Not Posted

8. Secondary Outcome: Percent Change in the 17-item Hamilton Depression (HAM-D17) Score From Baseline to 24 Weeks
Description: Evaluate the impact of GeneSight Psychotropic on response to psychotropic treatment as judged by the mean percent change in the 17-item Hamilton Depression (HAM-D17) score from baseline to end of Week 24 of the study. Scores range from 0 to 50, and lower scores are better outcomes. Percent change is defined as (week 24 score -baseline score) / (baseline score) x 100.
Time Frame: Baseline to week 24 visits
Population: Per Protocol - Due to unblinding before week 12 there was no longer a treatment as usual and guided treatment arm and it was pre-specified in the Protocol to include only the GeneSight Psychotropic Tested Arm/Group for this Outcome Measure
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | GeneSight Psychotropic Tested
Number analyzed (Participants) | 457
percentage of change | 42.5 (1.52)

9. Secondary Outcome: Percentage of Responders at Week 8 for QIDS-C16
Description: Adjusted percentage of responders at Week 8 in each treatment group on the 16-item Quick Inventory of Depression Symptomology (QIDS-C16). A responder is defined as a participant with at least 50% decrease from baseline in total scale score. Scores range from 0 to 27 with lower scores being better outcomes.
Time Frame: Week 8 visit info
Population: Intent-to-treat
Measure: Number; unit: percentage of subjects
Arm/Group | GeneSight Psychotropic Tested | Treatment As Usual
Number analyzed (Participants) | 677 | 621
percentage of subjects | 34.14 | 31.36
Statistical Analysis 1: Comparison: GeneSight Psychotropic Tested vs Treatment As Usual; Test type: Superiority; p = 0.2852, Generalized linear mixed model; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.90 to 1.43]

10. Secondary Outcome: Percentage of Responders at Week 8 for PHQ-9
Description: Adjusted percentage of responders at Week 8 in each treatment group on the 9-item Patient Health Questionnaire (PHQ-9). A responder is defined as a participant with at least 50% decrease from baseline in total scale score. Scores range from 0 to 27 with lower scores being better outcomes.
Time Frame: Week 8 visit info
Population: Intent-to-treat
Measure: Number; unit: percentage of subjects
Arm/Group | Treatment As Usual | GeneSight Psychotropic Tested
Number analyzed (Participants) | 676 | 620
percentage of subjects | 31.63 | 39.74
Statistical Analysis 1: Comparison: Treatment As Usual vs GeneSight Psychotropic Tested; Test type: Superiority; p = 0.0023, Generalized linear mixed model; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.43, 95% CI 2-sided [1.14 to 1.79]

11. Secondary Outcome: Percentage of Remitters at Week 12 Defined as QIDS-C16 ≤5
Description: as for outcome 4
Time Frame: week 12 visit info
Reporting Status: Not Posted

12. Secondary Outcome: Percentage of Remitters at Week 12 Defined as PHQ-9 <5
Description: as for outcome 4
Time Frame: week 12 visit info
Reporting Status: Not Posted

13. Secondary Outcome: Percentage of Remitters at Week 12 Defined as CGI-S ≤1
Description: as for outcome 4
Time Frame: week 12 visit info
Reporting Status: Not Posted

14. Secondary Outcome: Percentage of Responders at Week 12 for QIDS-C16
Description: as for outcome 4
Time Frame: Week 12 visit info
Reporting Status: Not Posted

15. Secondary Outcome: Percentage of Responders at Week 12 for PHQ-9
Description: as for outcome 4
Time Frame: Week 12 visit info
Reporting Status: Not Posted

16. Secondary Outcome: Percentage of Responders at Week 12 for CGI-S
Description: as for outcome 4
Time Frame: Week 12 visit info
Reporting Status: Not Posted

17. Secondary Outcome: Percentage of Responders at Week 12 for CGI-I
Description: as for outcome 4
Time Frame: Week 12 visit info
Reporting Status: Not Posted

18. Secondary Outcome: Percentage of Responders at Week 12 for CGI-EI
Description: as for outcome 4
Time Frame: Week 12 visit info
Reporting Status: Not Posted

19. Secondary Outcome: Percentage of Remitters at Week 8 Defined as QIDS-C16 ≤ 5 in Each Treatment Group
Description: Adjusted percentage of remitters at Week 8 in the 16-item Quick Inventory of Depression Symptomology (QIDS-C16) in each treatment group. A remitter is defined as a subject with a score ≤ 5. Scores range from 0 to 27 with lower scores being better outcomes.
Time Frame: week 8 visit info
Population: Intent-to-treat
Measure: Number; unit: percentage of subjects
Arm/Group | Treatment As Usual | GeneSight Psychotropic Tested
Number analyzed (Participants) | 677 | 621
percentage of subjects | 15.62 | 20.89
Statistical Analysis 1: Comparison: Treatment As Usual vs GeneSight Psychotropic Tested; Test type: Superiority; p = 0.0140, Generalized linear mixed model; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.43, 95% CI 2-sided [1.07 to 1.89]

20. Secondary Outcome: Percentage of Remitters at Week 8 Defined as PHQ-9 <5 in Each Treatment Group
Description: Adjusted percentage of remitters at Week 8 in each treatment group on the 9-item Patient Health Questionnaire (PHQ-9). A remitter is defined as a participant with score <5 on the PHQ-9. Scores range from 0 to 27 with lower scores being better outcomes.
Time Frame: week 8 visit info
Population: Intent-to-treat
Measure: Number; unit: percentage of subjects
Arm/Group | Treatment As Usual | GeneSight Psychotropic Tested
Number analyzed (Participants) | 677 | 620
percentage of subjects | 14.79 | 18.58
Statistical Analysis 1: Comparison: Treatment As Usual vs GeneSight Psychotropic Tested; Test type: Superiority; p = 0.0663, Generalized linear mixed model; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.98 to 1.76]

21. Secondary Outcome: Time to Response/Remission of Depressive Symptoms Over 12 Weeks;
Description: *Comment*: Time to response/remission is not an outcome measure that can accurately be reported from the way the data was collected. As specified in the updated SAP before the blind was broken, this was not analyzed and reported. Additionally, for patients in TAU, clinicians were blinded to the pharmacogenomic test result until after completion of the week 8 visit. Because unblinding may have occurred prior to week 12 assessments, data collected at week 12 were considered unblinded and are not reported.
Time Frame: week 4, 8, and 12 visit info
Reporting Status: Not Posted

22. Secondary Outcome: Percentage of Responders at Week 24 for HAM-D17 in the GeneSight Psychotropic Tested Treatment Group
Description: Adjusted percentage of responders at Week 24 in the GeneSight Psychotropic Tested treatment group on the 17-item Hamilton Depression Rating Scale (HAM-D17). A responder is defined as a participant with at least a 50% decrease from baseline in total scale score. Scores range from 0 to 50, and lower scores are better outcomes.
Time Frame: Baseline to week 24 visit info
Population: Per Protocol
Measure: Number; unit: percentage of subjects
Arm/Group | GeneSight Psychotropic Tested
Number analyzed (Participants) | 457
percentage of subjects | 44.3

23. Secondary Outcome: Percentage of Remitters at Week 24 Defined as HAM-D17 ≤7 in the GeneSight Psychotropic Tested Treatment Group
Description: Adjusted percentage of remitters at Week 8 defined as a score ≤7 in the 17-item Hamilton Depression Rating Scale (HAM-D17) in each treatment group. Scores range from 0 to 50, and lower scores are better outcomes.
  *Comment*: For patients in TAU, clinicians were blinded to the pharmacogenomic test result until after completion of the week 8 visit. Because unblinding may have occurred prior to week 12 assessments, all data collected at week 12 were considered unblinded and are not reported.
Time Frame: Baseline to week 24 visit info
Population: Per Protocol
Measure: Number; unit: percentage of subjects
Arm/Group | GeneSight Psychotropic Tested
Number analyzed (Participants) | 457
percentage of subjects | 31.1

24. Other Pre Specified Outcome: Generalized Anxiety Disorder 7-item (GAD-7) Scale
Description: The mean change in Generalized Anxiety Disorder 7-item (GAD-7) scale from week 12 to week 24
Time Frame: week 12 to week 24
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Generalized Anxiety Disorder 7-item (GAD-7) Scale
Description: The mean change in Generalized Anxiety Disorder 7-item (GAD-7) scale from baseline to week 8
Time Frame: baseline to week 8
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Generalized Anxiety Disorder 7-item (GAD-7) Scale
Description: The mean change in Generalized Anxiety Disorder 7-item (GAD-7) scale from baseline to week 12
Time Frame: baseline to week 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | GeneSight Psychotropic Tested | Treatment As Usual
All-Cause Mortality (participants affected / at risk) | 0/681 | 0/717
Serious Adverse Events (participants affected / at risk) | 3/681 | 2/717
Other Adverse Events (participants affected / at risk) | 0/681 | 0/717
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GeneSight Psychotropic Tested (N=681) | Treatment As Usual (N=717)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
transient hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
non cardiac chest pains (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-04-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT02109939/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT02109939/SAP_001.pdf